CLINICAL TRIAL: NCT02679404
Title: Sorin Universal REgistry on Aortic Valve Replacement
Acronym: SURE-AVR
Status: Terminated | Type: Observational
Why Stopped: Less data return than expected. The new Medical Device Regulation (MDR) implementation prompted the Sponsor to set up a broader scope post-market registry for all Corcym cardiovascular products (MANTRA).
Sponsor: Corcym S.r.l (Industry)
Responsible Party: Sponsor
Other Study IDs: APR001
Record Dates: First submitted 2016-01-27; First posted 2016-02-10 (Estimated); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Aortic Valve Disease; Aortic Stenosis
Keywords: Biological aortic valves; Mechanical aortic valves; Aortic conduits; Sutureless Aortic Valve
MeSH Terms: conditions — Aortic Valve Disease; Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Multi-center, International, Prospective, Non comparative, Non randomized, Open label.

5,000 patients to be enrolled approximately worldwide.

The objective of this registry is to collect safety and clinical performance post market data related to the procedure and follow-up of the Sorin Group aortic valve devices in accordance with the Instructions for Use (IFU).

This observational global registry is intended to collect data without requiring any deviation from the standard of care and IFU in each participating center. The participating centers shall include those patients that have provided their informed consent to participate in this registry in accordance with the local applicable regulations.

DETAILED DESCRIPTION:
SURE-AVR objective is to collect post market safety and performance data collected along the procedure and the relevant follow-up with Sorin Group aortic valve devices in accordance with the IFU to further evidence the safety and efficacy in a post-approval environment. All current and future Sorin Group aortic valve devices that have obtained CE-mark or other local regulatory and/or commercial approvals may be included in the registry. During the duration of the registry,other aortic valve replacement products or current devices might receive modifications and might become commercial available. This registry allows extensions for the inclusion of new products.

This observational global registry is intended to collect data without requiring any deviation from the standard of care and IFU in each participating center. The participating centers shall include those patients that have provided their informed consent to participate in this registry following the local applicable regulations.

The data collection shall be performed as per the local standard of care and without exposing the patient to any additional risk to the treatment (s)he would normally receive.

The registry is an open-ended project:

* Inclusions phase: open-ended
* Follow-up phase: annually throughout 5 years (7 and 10 years are optional).

The study shall be completed after the 10-year follow-up of the last patient.

ELIGIBILITY:
Inclusion Criteria:

* All patients must provide written or oral informed consent to participate in the registry depending on the local regulations.
* Patients having received a Sorin Group aortic valve device in accordance with the IFU

Exclusion Criteria: NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients having received a Sorin Group aortic valve device in accordance with the IFU can be included in the registry. Other than the indication and the contra-indications specified in each IFU, there are no specific inclusion and exclusion criteria since this registry has the aim to include all patients following "real life"/standard of care practices at participating centers. All patients must provide written or oral informed consent to participate in the registry following the local regulations.
Sampling Method: Probability Sample
Enrollment: 2758 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2021-03 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
Composite rate of valve related major adverse events (MAEs) | At 5 years follow-up
  To evaluate the composite rate of site reported valve related MAE defined as death, stroke and/or re-intervention (involving surgery or any other invasive therapy) at 5 years follow-up.

SECONDARY OUTCOMES:
Procedural timings | Intra-operative and at 30 days (average)
  Cross clamp time, intensive care unit and total length of hospital stay.
Clinical success | 30 days (average)
  The clinical success defined as a successful valve implantation without MAE at hospital discharge.
Improvement of clinical status | Annually through a 5-year follow-up, and 7 and 10-year follow-up in selected centers only.
  The improvement of clinical status defined as an improvement of at least one scale of the New York Heart Association (NYHA) classification between pre-procedure and annually throughout the duration of the registry.
Echocardiographic evaluation | Annually through a 5-year follow-up, and 7 and 10-year follow-up in selected centers only.
  Performance of the device in terms of hemodynamic behavior - Effective Orifice Area (cm²), Ejection Fraction (%),Mean Aortic Gradient (mmHg), Peak Aortic Gradient (mmHg), LV mass (g) - throughout the duration of the registry.
MAE during the duration of the registry | Annually through a 5-year follow-up, and 7 and 10-year follow-up in selected centers only.
  All site reported MAE rates during the duration of the registry.
Composite rate of valve related MAE | 4-year, and 7 and 10-year follow-up in selected centers only
  The composite rate of site reported valve-related MAE annually through a 4-year follow-up, and 7 and 10-year follow-up in selected centers only.
Valve-related Serious Adverse Event (SAE) | Annually through a 5-year follow-up, and 7 and 10-year follow-up in selected centers only.
  Other site reported valve-related SAE such as, but not limited to, bleeding, thromboembolism, valve thrombosis, endocarditis, non structural dysfunction, structural valve deterioration annually through a 5-year follow-up, and 7 and 10-year follow-up in selected centers only.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Gaggianesi, Study Director — Corcym S.r.l
Locations (52):
- United States (5):
  - Princeton Baptist Med Center, Birmingham, Alabama
  - River City Clinical Research, Jacksonville, Florida
  - Columbia University Hospital, New York, New York
  - Mount Carmel Hospital, Columbus, Ohio
  - Baylor Scott and White Research Institute, Plano, Texas
- Australia (2):
  - Melbourne Private Hospital, Melbourne
  - Royal Melbourne Hospital, Melbourne
- Hospital Salzburg, Salzburg, Austria
- Belgium (3):
  - UCL St Luc, Brussels
  - CHU Liège, Liège
  - CHR Namur, Namur
- Private cardiac center - Burgas, Burgas, Bulgaria
- Foothill Medical Centre - Calgary, Alberta, Calgary, Canada
- Czechia (2):
  - Center of Cardiovascular Surgery and Transplantation Brno, Brno
  - IKEM - Prague, Prague
- France (6):
  - CHU Bordeaux, Bordeaux
  - Clinique Saint Augustin, Bordeaux
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - Clinique la Protestante, Lyon
  - CHU La Timone, Marseille
  - CHU Rennes, Rennes
- Germany (2):
  - Universitätsklinikum Magdeburg, Magdeburg
  - Nuremberg Hospital, Nuremberg
- Sheba Medical Center, Tel Litwinsky, Israel
- Italy (12):
  - Azienda Ospedaliera Nazionale SS. Antonio e Biagio e C. Arrigo, Alessandria
  - Policlinico S.Orsola-Malpighi, Bologna
  - Fondazione Poliambulanza Istituto Ospedaliero, Brescia
  - Città di Lecce Hospital, Lecce
  - Fondazione Toscana Gabriele Monasterio-Presidio Ospedaliero di Massa, Massa
  - Centro Cardiologico Monzino, Milan
  - Istituto Clinico Sant'Ambrogio, Milan
  - Policlinico Paolo Giaccone, Palermo
  - IRCCS Policlinico San Donato, San Donato Milanese
  - Ospedale Ca' Foncello - Treviso, Treviso
  - Azienda Ospedaliero-Universitaria "Ospedali Riuniti" di Trieste, Trieste
  - Azienda Ospedaliero-Universitaria "S. Maria della Misericordia" di Udine, Udine
- Netherlands (2):
  - Amphia hospital Breda, Breda
  - UMC Groningen, Groningen
- National Heart Centre Singapore, Singapore, Singapore
- Vusch - Kosice, Košice, Slovakia
- Spain (4):
  - Hospital Juan Canalejo, A Coruña
  - Hospital Sant Pau, Barcelona
  - Hospital Reina Sofía, Córdoba
  - Hospital Clínico San Carlos, Madrid
- Switzerland (2):
  - University Hospital of Basel, Basel
  - Centre Hospitalier Universitaire Vaudois Lausanne, Lausanne
- United Kingdom (6):
  - Blackpool Teaching Hospital, Blackpool
  - Royal Sussex County Hospital - Brighton, Brighton
  - Bristol Royal Infirmary, Bristol
  - Hammersmith Hospital, London
  - King's College Hospital, London
  - Royal Brompton, London

IPD SHARING:
Plan to Share IPD: No